CLINICAL TRIAL: NCT03249623
Title: Weaning From Mechanical Ventilation: Comparison of Open-Loop Decision Support System and Routine Care, in the General Intensive Care Unit
Brief Title: Individualised Weaning From Mechanical Ventilation in General ICU
Acronym: iCareWean_CW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 226610; 2017-002627-25 (EudraCT Number)
Record Dates: First submitted 2017-06-22; First posted 2017-08-15 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Ventilatory Failure
Keywords: Weaning; Intensive Care; Individualised Care; Open-Loop Decision Support System; Respiratory Failure; Mechanical Ventilation; Spontaneous breathing Tests; Extubation
MeSH Terms: conditions — Hypoventilation; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: After randomisation, for patients randomised in the Beacon group, the Beacon system will actively advice clinicians on ventilatory settings to adapt the ventilator to patient's individual clinical situation and corresponding clinical intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Beacon Caresystem (Experimental): On randomisation to the Beacon group, a Beacon Caresystem will be connected to the patient. This involves connecting a pulse oximeter to the patient's finger (toe or ear) to measure pulse oximetry oxygen saturation and pulse, and placing a standard clinical respiratory gas analysis and flow sensor in the respiratory tubing connecting the ventilator to the patient. This sensor allows measurement of respiratory pressure, flow and volume; plus respiratory gas CO2 and O2.
  Interventions: Device: Beacon Caresystem
- Standard Care (No Intervention): For this group mechanical ventilation is managed according to standard care. A Beacon CareSystem will be connected to the patient, as for the Beacon Randomisation group, but the system will be used solely for data collection, and advice will be disabled. Physiological variables captured in this arm of the study will mirror the intervention arm. Decision relating to weaning, extubation, reintubation and sedation including level of seniority of personnel involved in the decision tree process will be documented accordingly.

INTERVENTIONS:
Device: Beacon Caresystem — The core of the system is a set of physiological models including pulmonary gas exchange, acid-base chemistry, lung mechanics, and respiratory drive. The Beacon Caresystem tunes these models to the individual patient such that they describe accurately current measurements. Once tuned, the models are used by the system to simulate the effects of changing ventilator settings. The results of these simulations are then used calculate the clinical benefit of changing ventilator settings by balancing the competing goals of mechanical ventilation.
  Arms: Beacon Caresystem

SUMMARY:
Patients residing in the intensive care unit typically receive mechanical ventilatory support. Selecting the appropriate level of mechanical ventilation is not trivial, and it has been shown that lung protective settings can reduce mortality in patients with lung injury. Despite being a life- saving therapy, duration of mechanical ventilation should be kept at a minimum to reduce effects of immobilization, long-term sedation, patient discomfort, risk of ventilator associated pneumonia, leading to decreasing mortality and economic costs etc. The duration of mechanical ventilation is also an important factor in weaning from ventilatory support, with prolonged ventilator support making the weaning process more difficult.

The purpose of this study is to compare mechanical ventilation following advice from the Beacon Caresystem to that of standard care in general medical intensive care unit (ICU) patients, from the start of requiring invasive mechanical ventilation until successful extubation. The Beacon Caresystem will be compared to standard care to investigate whether use of the system results in similar care or reduced time for weaning from mechanical ventilation.

DETAILED DESCRIPTION:
All patients admitted to the ICU with mechanical ventilation are screened for inclusion. Patients receiving invasive mechanical ventilation (≥ 24 h) will be considered for inclusion in the study on a daily basis. Patient screening will be performed by clinical researchers or a delegated clinician and consent/assent will be sought. Then patients will be randomised to the Beacon group or Standard Care group. Randomisation will be performed using sealed envelopes, and in blocks of patients, allowing interim analysis of results in appropriate steps during the study. To avoid that results are affected by patient disease type, randomisation will be stratified for equal distribution between randomisation groups.

Patients will be randomly assigned to either standard care of mechanical ventilation, or to follow the advice of the Beacon Caresystem. The results of these two strategies will then be compared based upon the following outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patient is expected to be on invasive mechanical ventilation more 24 hours.
* Age > 18 years
* Haemodynamically stable (with instability defined by the presence of two or more of the following criteria: acidosis pH < 7.2, poor urine output < 0.5ml/kg, use of vasopressors, e.g. noradrenline > 25 μg/min).
* Patient consent or, in the case that the patient is unable, assent from the next of kin or treating physician following understanding and accept of oral and written information describing the study

Exclusion Criteria:

* The absence of an arterial catheter for blood sampling at study start.
* Medical history of home mechanical ventilation which may lead to prolonged stay in the ICU, including long term oxygen therapy and non-invasive ventilation not associated with sleep apnoa.
* Clinical conditions requiring treatment with extracorporeal membrane oxygenation, i.e. an inspired oxygen of 100% for more than 24 hours.
* Head trauma or other conditions where intra-cranial pressure may be elevated and tight regulation of arterial CO2 level is paramount.
* Primary neurological patients (Glasgow coma score <10, neurologic damage with limited prognosis, stroke hemiplegia).
* Severe heart failure, classified as grade 4 of the Association of Cardiology guidelines [2].
* End stage liver disease.
* Multiple medical ICU admissions, i.e. more than one admission.
* Corrective orthognathic surgery.
* Esophageal surgery.
* Morbidly obese patients defined as either BMI>45, or 35<BMI<45 with APACHEII score on admission greater than 24.
* Pregnancy.
* Mechanical ventilation initiated for more for 24 hours in other centers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Length of mechanical ventilation | Daily assessment of requirement of mechanical ventilation from the time of randomisation until the date of liberation from mechanical ventilation, up to 12 months.
  Length of mechanical ventilation, defined as either the time of intubation in the ICU, or the time of admission to the ICU following previous intubation for surgery, and until successful extubation, with successful

SECONDARY OUTCOMES:
Time to spontaneous ventilation | Daily assessment of spontaneous ventilation from the date of randomisation until the date the patient starts breathing spontaneously, up to 12 months.
  It is defined as the time taken to wean from mandatory mode of ventilation
Time to extubation | Daily assessment of time to extubation from the date of initiation of spontaneous ventilation until the date of liberation from mechanical ventilation, up to 12 months.
  It is defined as the time the decision is made to proceed with removal of the endotracheal tube or tracheal decannulation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela P Vizcaychipi, MD PhD FFICM, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- The Magill Department of Anaesthesia, Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rees SE, Karbing DS. Determining the appropriate model complexity for patient-specific advice on mechanical ventilation. Biomed Tech (Berl). 2017 Apr 1;62(2):183-198. doi: 10.1515/bmt-2016-0061. PMID 27930361
- [Result] Rees SE, Karbing DS. Model-based advice for mechanical ventilation: From research (INVENT) to product (Beacon Caresystem). Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:5331-4. doi: 10.1109/EMBC.2015.7319595. PMID 26737495
- [Result] Weinreich UM, Thomsen LP, Rees SE, Rasmussen BS. The effects of oxygen induced pulmonary vasoconstriction on bedside measurement of pulmonary gas exchange. J Clin Monit Comput. 2016 Apr;30(2):207-14. doi: 10.1007/s10877-015-9703-x. Epub 2015 May 12. PMID 25962614
- [Derived] Vizcaychipi MP, Karbing DS, Martins L, Gupta A, Moreno-Cuesta J, Naik M, Welters I, Singh S, Randell G, Osman L, Rees SE. Evaluation of decision support to wean patients from mechanical ventilation in intensive care: a prospective study reporting clinical and physiological outcomes. J Clin Monit Comput. 2025 Apr;39(2):393-404. doi: 10.1007/s10877-024-01231-5. Epub 2024 Nov 9. PMID 39520605
- [Derived] Vizcaychipi MP, Martins L, White JR, Karbing DS, Gupta A, Singh S, Osman L, Moreno-Cuesta J, Rees S. Intensive Care Weaning (iCareWean) protocol on weaning from mechanical ventilation: a single-blinded multicentre randomised control trial comparing an open-loop decision support system and routine care, in the general intensive care unit. BMJ Open. 2020 Sep 2;10(9):e042145. doi: 10.1136/bmjopen-2020-042145. PMID 32878764
- See also: Details of the Beacon System — http://mermaidcare.com
- See also: Sponsor website — http://www.chelwest.nhs.uk